CLINICAL TRIAL: NCT01930396
Title: Intermittent HEMOdialysis Anticoagulation With TINzaparin Versus Unfractionated Heparin: A Pilot Multicentre Randomized Controlled Trial (HEMO-TIN Trial)
Brief Title: Use of Tinzaparin for Anticoagulation in Hemodialysis
Acronym: HEMO-TIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christine Ribic (Other)
Collaborators: McMaster University (Other); LEO Pharma (Industry)
Responsible Party: Sponsor-Investigator, Christine Ribic, Nephrologist, St. Joseph's Healthcare Hamilton
Organization: St. Joseph's Healthcare Hamilton (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-7822377
Record Dates: First submitted 2013-08-22; First posted 2013-08-28 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Failure, Chronic
Keywords: Hemodialysis; Anticoagulation; Tinzaparin; Unfractionated Heparin; Randomized Controlled Trial
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tinzaparin; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tinzaparin (Experimental)
  Interventions: Drug: Tinzaparin; Drug: Placebo (for Unfractionated Heparin)
- Unfractionated Heparin (Active Comparator)
  Interventions: Drug: Unfractionated Heparin; Drug: Placebo (for Tinzaparin)

INTERVENTIONS:
Drug: Tinzaparin
  Other Names: Innohep
  Arms: Tinzaparin
Drug: Unfractionated Heparin
  Other Names: Heparin LEO
  Arms: Unfractionated Heparin
Drug: Placebo (for Tinzaparin) — 0.9% Normal Saline
  Arms: Unfractionated Heparin
Drug: Placebo (for Unfractionated Heparin) — 0.9% Normal Saline
  Arms: Tinzaparin

SUMMARY:
The HEMO-TIN trial is designed to look at both the safety (bleeding risk) and effectiveness (clotting risk) of tinzaparin compared with unfractionated heparin for anticoagulation in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* End stage renal disease maintained on outpatient hemodialysis for >= 3 months
* Frequency of hemodialysis: 3 times per week
* Anticoagulation with an unfractionated heparin protocol for at least 4 weeks
* Patient or legal guardian able to provide written consent
* Baseline INR <= 1.3
* Baseline platelet count >= 80,000 x 10^9/L

Exclusion Criteria:

* Therapeutic systemic anticoagulation
* Clinically apparent bleeding in the last 2 months
* High risk of bleeding
* Planned major surgery in the next 4 months
* Major surgery in the past 48 hours
* Pregnant or lactating
* Child bearing potential
* Allergy/intolerance to heparin or history of heparin induced thrombocytopenia
* Current participation in a related randomized drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of major, clinically important non-major or minor bleeding | 26 weeks

SECONDARY OUTCOMES:
Clotting in extracorporeal dialysis circuit | During Hemodialysis (weekly for 26 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christine M Ribic, MD, MSc, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593